CLINICAL TRIAL: NCT03347474
Title: Deep Brain Stimulation of Nucleus Accumbens for Methamphetamine Addiction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of the Department of Functional Neurosurgery, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-10-25 DBS-NAc Meth
Record Dates: First submitted 2017-09-03; First posted 2017-11-20 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Treatment Methamphetamine Addiction
Keywords: Bilateral Nucleus Accumbens; Methamphetamine Addiction

STUDY DESIGN:
Intervention Model Description: All subjects will receive bilateral surgical implantation of DBS system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral surgical implantation of DBS system to NAc (Experimental)
  Interventions: Procedure: Bilateral surgical implantation of DBS system to NAc

INTERVENTIONS:
Procedure: Bilateral surgical implantation of DBS system to NAc — The Medtronic, PINS and SceneRay DBS device will be utilized in the present study.

SUMMARY:
The main objective of this study is to assess the efficacy of bilateral deep brain stimulation (DBS) of the Nucleus Accumbens(NAc) as a novel treatment in severe methamphetamine addiction. Our hypothesis is that bilateral DBS of the NAc will significantly reduce the craving for methamphetamine.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR diagnosis of Drug addiction disorder;
* Age 18-65 years old;
* Proficiency in Mandarin language;
* Failure to detox more than three times;
* Capacity to provide informed consent (understanding of the study purpose and methods);

Exclusion Criteria:

* Multidrug abuse and formation of addiction;
* Serious and unstable organic diseases (e.g. unstable coronal heart disease);
* Any history of seizure disorder or hemorrhagic stroke;
* Past stereotactic neurosurgical intervention;
* Neurological disease (Abnormal PET-CT, MRI, EEG)
* Contraindications of MRI-examination, e.g. implanted cardiac pacemaker/ heart defibrillator;
* Contraindications of stereotactic intervention, e.g. increased bleeding disposition, cerebrovascular diseases (e.g. arteriovenous malfunction, aneurysms, systemic vascular diseases);
* HIV positive;
* Pregnancy and/or lactation;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
change in 10-point visual analog scale of carving | Baseline (preoperative),3 months,6 months, 12 months
  The score of scale is from 0 to 10. 0 represents no carving for drug, 10 means the greatest degree of carving for drug.
change in Obsessive Compulsive Drug Use Scale | Baseline (preoperative),3 months,6 months, 12 months

SECONDARY OUTCOMES:
Side Effect | Baseline（preoperative）,3 months, 6 months, 12months
Change in the Hamilton Anxiety Scale | Baseline（preoperative）,3 months, 6 months, 12months
Change in the Hamilton Depression Scale | Baseline（preoperative）,3 months, 6 months, 12 months
Change in the Quality of Life Assessment (SF-36) | Baseline（preoperative）,3 months, 6 months, 12 months
Change in World Health Organization Quality of Life-BREF(WHO-BREF) | Baseline（preoperative）,3 months,6 months, 12 months
Chang in Pittsburgh Sleep Quality Index | Baseline（preoperative）,3 months,6 months, 12 months
Neuropsychological measures(Scores of cognitive battery) | Baseline（preoperative）,6 months,12 months
Change in Fagerstrom Test of Nicotine Dependence(FTND) | Baseline（preoperative）,3 months,6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital Functional Neurosurgery, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Kuhn J, Moller M, Treppmann JF, Bartsch C, Lenartz D, Gruendler TO, Maarouf M, Brosig A, Barnikol UB, Klosterkotter J, Sturm V. Deep brain stimulation of the nucleus accumbens and its usefulness in severe opioid addiction. Mol Psychiatry. 2014 Feb;19(2):145-6. doi: 10.1038/mp.2012.196. Epub 2013 Jan 22. No abstract available. PMID 23337942